CLINICAL TRIAL: NCT02626494
Title: Neurobiological Adaptations and Pharmacological Interventions in Cocaine Addiction: The Role of Glutamate
Brief Title: Neurobiological Adaptations and Pharmacological Interventions in Cocaine Addiction
Acronym: CoGlu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Collaborators: Zurich Center for Integrative Human Physiology (Other); Swiss Federal Institute of Technology (Other); Max-Planck-Institut Tübingen (Unknown)
Responsible Party: Principal Investigator, Dr. med. Marcus Herdener, Dr. med Marcus Herdener, Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CoGlu_PUK_ZH_2014_0010
Record Dates: First submitted 2015-05-20; First posted 2015-12-10 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Cocaine Addiction
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cocaine Group (Experimental): n-AC and placebo will be given according to a double-blind, placebo-controlled cross-over design. Subjects receive 4 doses of n-AC/placebo over 2 consecutive days (total dose=4800mg; individual dose=1200mg). Subjects will take the first 2 doses of n-AC/placebo 5 days after the screening assessment (one in the morning, one in the evening), and the last 2 dose 1h prior to scanning, with 12 hours dosing intervals in between. 14 days later n-AC/placebo will be administered analogously as described above. Preparation and blinding of n-AC and placebo capsules will be performed by the Kantonsapotheke Zürich according to the guidelines of Good Manufacturing Practice.
  Interventions: Drug: N-Acetylcystein; Drug: Placebo
- Healthy Control Group (Active Comparator): n-AC and placebo will be given according to a double-blind, placebo-controlled cross-over design. Subjects receive 4 doses of n-AC/placebo over 2 consecutive days (total dose=4800mg; individual dose=1200mg). Subjects will take the first 2 doses of n-AC/placebo 5 days after the screening assessment (one in the morning, one in the evening), and the last 2 dose 1h prior to scanning, with 12 hours dosing intervals in between. 14 days later n-AC/placebo will be administered analogously as described above. Preparation and blinding of n-AC and placebo capsules will be performed by the Kantonsapotheke Zürich according to the guidelines of Good Manufacturing Practice.
  Interventions: Drug: N-Acetylcystein; Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcystein — n-AC will be given according to a double-blind, placebo-controlled cross-over design. Subjects receive 3 doses of n-AC over 2 consecutive days (total dose=4800mg; individual doses=2x1200mg, 1x2400mg). Subjects will take 2 first doses (à 1200mg) of n-AC 5 days after the screening assessment (one in the morning, one in the evening), and the last dose (2400mg) 1h prior to scanning, with 12 hours dosing intervals in between. Preparation and blinding of n-AC capsules will be performed by the Kantonsapotheke Zürich according to the guidelines of Good Manufacturing Practice.
Drug: Placebo — 14 days before or after, placebo will be administered analogously as described with n-AC. Placebo will be given according to a double-blind, placebo-controlled cross-over design. Subjects receive 3 doses of placebo over 2 consecutive days (total dose=4800mg; individual doses=2x1200mg, 1x2400mg). Subjects will take 2 first doses (à 1200mg) of placebo 1 day before scanning (one in the morning, one in the evening), and the last dose (2400mg) 1h prior to scanning, with 12 hours dosing intervals in between. Preparation and blinding of placebo capsules will be performed by the Kantonsapotheke Zürich according to the guidelines of Good Manufacturing Practice.

SUMMARY:
This study aims at testing for the impact of glutamatergic changes on drug craving in cocaine addiction, and to evaluate the effects of n-acetylcysteine (n-AC) on both glutamate homeostasis and craving using a randomized, double-blind, placebo controlled cross-over design.

DETAILED DESCRIPTION:
Cocaine addiction is a devastating disorder with potentially harmful psychological, physical and social consequences. Despite its clinical importance, there is currently no approved pharmacological treatment available for cocaine addiction. However, preclinical research has recently identified potentially promising targets for pharmacotherapeutic approaches mainly based on advances in the understanding of neuroplastic alterations associated with repeated cocaine administration in animals.

Preclinical animal models revealed that chronic administration of cocaine leads to decreased basal levels of glutamate within the nucleus accumbens a key region of the neural reward circuitry; in turn, the reinstatement of drug seeking results in enhanced glutamatergic transmission. However, little is known about similar changes in humans, and about their functional role for addictive behavior, mainly due to methodological restrictions. The investigators thus aim to examine the changes associated with chronic cocaine use on glutamate homeostasis in humans using a newly developed proton magnetic resonance spectroscopy (1H-MRS) protocol. This method allows for the quantification of brain metabolites such as glutamate in specific regions of the human brain even within small subcortical volumes of interest such as the nucleus accumbens that have been hitherto difficult to assess.

Interestingly, the administration of n-AC restored the glutamate homeostasis in rats and reduced their drug reinstatement behavior. Therefore, the present study aims at investigating if a pharmacological challenge of n-AC influences glutamate homeostasis in humans and whether these possible modulations are linked to cocaine craving.

Power analyses to identify the sample size of this study, were done with a focus on 1H-MRS, the most critical procedure in this context within our project. Assuming a mean conservative effect size of d=0.80, an α-error probability of 5%, and a conservative power estimation of 80% and considering a drop-out rate of about 30%, investigators plan to measure 30 cocaine dependent patients and 30 healthy controls.

Imaging data of low quality (e.g. due to movement artifacts) will be excluded. If imaging data has to be excluded or if participants do not finish the experiment, the investigators will additionally recruit more participants in order to assess the planned sample size.

Throughout the duration of the entire study, the conductance of pre-defined key processes will constantly be monitored by an independent monitor in specified visit intervals to ensure that the study is conducted in accordance with the approved protocol, good clinical practice, and the applicable regulatory requirement in order to protect the rights and well-being of study participants and integrity of data.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine use disorder vs. no substance use
* Magnetic resonance imaging compatibility

Exclusion Criteria:

* Regular use of other psychoactive drugs
* Comorbidity of other psychiatric disorders
* Neurological or somatic disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Glutamatergic alterations in cocaine users assessed by 1H-MRS as glutamate concentrations in the nucleus accumbens expressed as glutamate ratios in relation to water [glutamate/water] | It will be assessed in the placebo condition at either the 1.measurement (approximately 1.5h after ingestion of the last dose), on average 2 days after the initial assessment of the subject or at the 2.measurement (in average 14 days after 1.measurement)
  - Changes in basal glutamatergic neurotransmission in the nucleus accumbens in cocaine addiction will be assessed via 1H-MRS.
Impact of n-acetylcystein on glutamate homeostasis assessed by 1H-MRS as glutamtate concentrations in the nucleus accumbens expressed as glutamate ratios in relation to water [glutamate/water] | The impact of n-AC will be assessed by comparing n-AC and placebo condition, with an average time interval of 14 days between measurements.
  * The impact of n-AC on glutamatergic neurotransmission in cocaine addiction will be assessed via 1H-MRS.
Impact of n-acetylcystein on craving assessed by visual analog scales | The impact of n-AC will be assessed by comparing n-AC and placebo condition with an average time interval of 2 weeks between measurements.
  * Craving will be assessed via subjective ratings on visual analog scales
  * The impact of n-AC will be assessed by comparing craving in cocaine dependent individuals under n-AC and placebo.

SECONDARY OUTCOMES:
Alterations in frontostriatal networks indicated by connectivity coefficients assessed by functional magnetic resonance imaging | Alterations in frontostriatal will be assessed by comparing n-AC and placebo condition with an average time interval of 2 weeks.
  * Alterations in frontostriatal networks will be assessed via magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Herdener, MD, Principal Investigator — Center for Addicitve Disorders
Locations (1):
- Psychiatric University Hospital, Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Engeli EJE, Preller KH, Rieser NM, Klar J, Staempfli P, Hulka LM, Kirschner M, Seifritz E, Herdener M. N-acetylcysteine reduces prefrontal reactivity to cocaine cues in individuals with cocaine use disorder. Front Psychiatry. 2025 Feb 27;15:1489194. doi: 10.3389/fpsyt.2024.1489194. eCollection 2024. PMID 40083914